CLINICAL TRIAL: NCT02077205
Title: Manualised Cognitive Behavioral Therapy of Anxiety Disorders in Children and Adolescents in Routine Care Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Prof. Dr. Silvia Schneider, Prof. Dr., Ruhr University of Bochum
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: no funding
Record Dates: First submitted 2014-02-04; First posted 2014-03-04 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-02

CONDITIONS: Anxiety Disorders
Keywords: Diagnostic and Statistical Manual of Mental Disorders-IV/-5: Anxiety Disorders in children
MeSH Terms: conditions — Anxiety Disorders; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Manualised Cognitive Behavioral Therapy (Experimental): Manualised Cognitive Behavioral Therapy in a Routine Care Setting
  Interventions: Behavioral: Manualised Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Manualised Cognitive Behavioral Therapy — 16 Sessions of Manualised Cognitive Behavioral Therapy in a Routine Care Setting

SUMMARY:
Manualised Cognitive Behavioral Therapy for children and adolescents with anxiety disorders is evaluated in a routine care setting to evaluate the efficacy of the intervention. Children and adolescents receive manualized Cognitive Behavioral Therapy for anxiety disorder.

It is expected, that the intervention will result in less anxiety / lower scores on the primary and secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 4-18 years
* Primary diagnosis of an anxiety disorder:

  1. Generalized Anxiety Disorder
  2. Social Phobia
  3. Separation Anxiety Disorder
  4. Panic Disorder +/- Agoraphobia
  5. Specific Phobia

Exclusion Criteria:

* Other primary diagnoses
* Significant intellectual impairment

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Severity rating of diagnosis (according to the Kinder-DIPS) | Changes in severity rating from pre- to post-assessment (post-assessment takes place 30 weeks after the pre-assessment on average) and to 6-month-follow-up (which takes place about 6 months after the post-assessment)
Spence Children's Anxiety Scale (SCAS) | Changes on the SCAS from pre- to post-assessment (post-assessment takes place 30 weeks after the pre-assessment on average) and to 6-month-follow-up (which takes place about 6 months after the post-assessment)
Clinical Global Improvement Impression (CGI-I) | Changes on the CGI-I from post-assessment (post-assessment takes place 30 weeks after the pre-assessment on average) to 6-month-follow-up (which takes place about 6 months after the post-assessment)
Interference rating as assessed by the "Beurteilung der Beeinträchtigung/ Einschränkung des Patienten" (BEE) | Changes in interference rating from pre- to post-assessment (post-assessment takes place 30 weeks after the pre-assessment on average) and to 6-month-follow-up (which takes place about 6 months after the post-assessment)
  The German questionnaire "Beurteilung der Beeinträchtigung/ Einschränkung des Patienten" (BEE) assesses the degree of interference.

SECONDARY OUTCOMES:
Depression as measured by the Short Moods and Feelings Questionnaire (SMFQ) | Changes in the SMFQ from pre- to post-assessment (post-assessment takes place 30 weeks after the pre-assessment on average) and to 6-month-follow-up (which takes place about 6 months after the post-assessment)
Strengths and Difficulties Questionnaire (SDQ) | Changes on the SDQ from pre- to post-assessment (post-assessment takes place 30 weeks after the pre-assessment on average) and to 6-month-follow-up (which takes place about 6 months after the post-assessment)

CONTACTS AND LOCATIONS:
Locations (1):
- Ruhr-University of Bochum, Department of Psychology, AE Klinische Kinder- und Jugendpsychologie, Bochum, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Krause K, Zhang XC, Schneider S. Long-Term Effectiveness of Cognitive Behavioral Therapy in Routine Outpatient Care for Youth with Anxiety Disorders. Psychother Psychosom. 2024;93(3):181-190. doi: 10.1159/000537932. Epub 2024 Apr 12. PMID 38615662